CLINICAL TRIAL: NCT06258902
Title: Odevixibat Pregnancy and Lactation Surveillance Program: A Post-marketing, Long-term, Observational, Descriptive Study to Assess the Risk of Pregnancy and Maternal Complications and Adverse Effects on the Developing Fetus, Neonate, and Infant Among Individuals Exposed to Odevixibat During Pregnancy and/or Lactation
Brief Title: Odevixibat Pregnancy and Lactation Surveillance Program: A Study to Evaluate the Safety of Odevixibat During Pregnancy and/or Lactation
Status: Recruiting | Type: Observational
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Other Study IDs: A4250-017
Record Dates: First submitted 2024-02-02; First posted 2024-02-14 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Pregnancy Related
Keywords: Rare disease; PFIC; Pregnancy; Lactation
MeSH Terms: conditions — Rare Diseases; Breast Feeding

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The participants of this study will be of any age who are exposed to at least 1 dose of odevixibat at any time during pregnancy (from 1 day prior to conception to pregnancy outcome) and/or at any time during lactation (up to 12 months of infant age or weaning, whichever comes first.

This study will collect data obtained via a variety of sources, including enrolled pregnant or lactating participants, the healthcare providers (HCP) involved in their care or the care of their infants, if applicable, and Albireo pharmacovigilance.

Study start date is either start of data collection or first patient enrolled whatever occurs earlier.

The surveillance program is strictly observational; the schedule of office visits and all treatment regimens are determined by HCPs. Only data that are routinely documented in patients' medical records as part of usual care will be collected.

No additional laboratory tests or HCP assessments will be required as part of this surveillance program.

ELIGIBILITY:
Inclusion Criteria:

* Exposure to at least 1 dose of odevixibat at any time during pregnancy (from 1 day prior to conception to pregnancy outcome) and/or at any time during lactation (up to 12 months of infant age or weaning, whichever comes first).
* Informed consent or IRB-/EC-approved waiver of informed consent (not applicable if reported by Albireo PV according to usual pharmacovigilance practices)

Exclusion Criteria:

* Refusal to provide informed consent, if required

Sex: Female
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Child-bearing potential women: individuals of any age who are exposed to at least 1 dose of odevixibat at any time during pregnancy and/or lactation.
Study Population: The main population will be individuals of any age who are exposed to at least 1 dose of odevixibat at any time during pregnancy (from 1 day prior to conception to pregnancy outcome) and/or at any time during lactation (up to 12 months of infant age or weaning, whichever comes first).
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2023-09-28 (Actual); Primary Completion 2032-05-31 (Estimated); Study Completion 2032-05-31 (Estimated)

PRIMARY OUTCOMES:
Prevalence rate of major congenital malformations (MCM) at birth | At birth
  An abnormality of body structure or function that is present at birth; is of prenatal origin (i.e. birth defect); has significant medical, social or cosmetic consequences for the affected individual; and typically requires medical intervention.

SECONDARY OUTCOMES:
Prevalence rate of minor congenital malformations at birth | At birth
Prevalence rate of molar or ectopic pregnancy | Throughout pregnancy, an average of 9 months
  Molar pregnancy is defined as an abnormal pregnancy that happens when a sperm fertilizes an egg that does not contain any genetic material. Ectopic pregnancy is defined as a pregnancy that occurs outside of the uterine cavity, usually in one of the fallopian tubes.
Prevalence rate of fetal loss | Throughout pregnancy, an average of 9 months
  A fetal loss that occurs for any reason at any time during pregnancy. This includes spontaneous abortion (SAB), stillbirth, elective or therapeutic abortion, fetal loss (type not specified).
Prevalence rate of live birth | At birth
  The birth of a living fetus at ≥ 20 gestational weeks or, if gestational age is unknown, weighing ≥ 350g.
Prevalence rate of preterm birth | At birth
Prevalence rate of small for gestational age (SGA) | At birth
  Birth weight <10th percentile for sex and gestational age using standard growth charts for full and preterm live-born infants.
Prevalence rate of neonatal death | Within the first 28 days of life
Prevalence rate of infant death | Throughout the first year of life
Prevalence rate of postnatal growth deficiency | Throughout the first year of life
  Weight, length or head circumference in <10th percentile for sex and age using standard growth charts.
Prevalence rate of infant developmental delay | Throughout the first year of life
  Failure to achieve the developmental milestones for chronological age, as defined by the Centers for Disease Control and Prevention (CDC)
Prevalence rate of infant hospitalization due to serious illness | Throughout the first year of life
  Infant hospital visit due to a serious (i.e. results in significant disability, incapacity, or death; is life-threatening; requires inpatient or prolonged hospitalization; or is considered medically important)

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (1):
- Virtual Research Coordination Center Odevixibat (BYLVAY) Pregnancy Surveillance Program, Wilmington, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, annotated case report form, statistical analysis plan, and dataset specifications.
  Patient level data will be anonymized and study documents will be redacted to protect the privacy of study participants.
Time Frame: Where applicable, data from eligible studies are available 6 months after the studied medicine and indication have been approved in the US and/or EU.
Access Criteria: Further details on Ipsen's sharing criteria and process for sharing are available here (https://www.ipsen.com/science/clinical-trials/clinical-data-transparency/).
URL: https://www.ipsen.com/science/clinical-trials/clinical-data-transparency/